CLINICAL TRIAL: NCT07328373
Title: Neurobiological and Genomic Predictors of Relapse After Discontinuation of Antidepressant Treatment in Major Depressive Disorder: An Observational Prospective Study
Brief Title: Neurobiological and Genomic Predictors of Relapse in Depression
Acronym: MDD
Status: Recruiting | Type: Observational
Sponsor: Mehmet Kemal Arikan (Other)
Responsible Party: Sponsor-Investigator, Mehmet Kemal Arikan, Professor Doctor, Uskudar University
Organization: Uskudar University (Other)
Other Study IDs: WSM_MDD
Record Dates: First submitted 2025-12-02; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Healthy; Major Depressive Disorder (MDD)
Keywords: Quantitative EEG; Rapid Eye Movement; Sleep EEG; Event Related Potential; P300; Alpha Asymmetry; Oddball Paradigm; relapse; recurrence; antidepressants; dna; rna; epigenetic; ssri; snri; methylation; quality of life; stress; magnetic resonance imaging; diffusion tensor imaging
MeSH Terms: conditions — Depressive Disorder, Major; Recurrence | interventions — Selective Serotonin Reuptake Inhibitors; Paroxetine; Fluoxetine; Sertraline; Escitalopram; Duloxetine Hydrochloride; Venlafaxine Hydrochloride; Antidepressive Agents, Second-Generation; Bupropion; Mirtazapine; Trazodone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood will be retained for DNA, RNA, microRNA extraction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Depression-Relapsed Prospectively Followed: This cohort includes patients whose long-term outcome is unknown at the start of the study. They are enrolled, treated, and monitored over time. At the study's conclusion, they will be retrospectively categorized as "Relapsers".
  Interventions: Drug: Antidepressant Medications
- Healthy Control: This group is composed of individuals with no history of psychiatric illness. Data is collected at a single time point to establish a healthy baseline for all biomarkers.
- Recurrent Depression Retrospectively Defined: Group A (Retrospective / Known Phenotype): This group consists of patients with a confirmed history of recurrent depression. Recurrence defined as no relapse within 1 year after discontinuation of medication. Data for this group is collected at a single time point (Baseline/T0).
  Interventions: Drug: Antidepressant Medications
- Non-Recurrent Depression Retrospectively Defined: This group consists of patients with a confirmed history of a single depressive episode or no relapse within 1 year after discontinuation of medication. Data for this group is collected at a single time point (Baseline/T0).
- Depression-Non-Relapsers Prospectively Followed: This cohort includes patients whose long-term outcome is unknown at the start of the study. They are enrolled, treated, and monitored over time. At the study's conclusion, they will be retrospectively "Non-Relapsers" (in Remission).
  Interventions: Drug: Antidepressant Medications

INTERVENTIONS:
Drug: Antidepressant Medications — Second generation antidepressants under "selective serotonin reuptake inhibitor" group
  Other Names: Selective Serotonin Reuptake Inhibitors, e.g., paroxetine, fluoxetine, sertraline, escitalopram; Selective Norepinephrine Reuptake Inhibitors, e.g., duloxetine, venlafaxine; Atypical Antidepressants, e.g., bupropion, mirtazapine, trazodone
  Groups: Depression-Non-Relapsers Prospectively Followed; Depression-Relapsed Prospectively Followed; Recurrent Depression Retrospectively Defined

SUMMARY:
The goal of this observational study is to test whether the discontinuation of antidepressant medications for patients with depression can be decided after the normalization of biological parameters. The main questions it aims are:

1. When patients with depression treated with antidepressants, does their brain activity also become normal? If so,
2. Then, can we stop the antidepressant treatment and expect minimum repeat of depression?

The participants who receive a specific antidepressant treatment will be asked to:

* Undergo quantitative electroencephalography (qEEG),
* Record Event-related potential (ERP),
* Record Sleep EEG
* Answer Hamilton Depression Rating Scale question their psychiatrists asked
* Give blood sample for genetic analysis
* Repeat the above mentioned procedures for at least 3 times during their treatment period.

Researchers will compare the results of patients with the results of healthy controls.

DETAILED DESCRIPTION:
When Should Antidepressant Treatment Be Discontinued? A Prospective Healthy-Controlled Case-Control Study

Background First-line treatments for Major Depressive Disorder (MDD) include second-generation antidepressants-such as selective serotonin reuptake inhibitors (SSRIs) and serotonin-norepinephrine reuptake inhibitors (SNRIs)-and/or evidence-based psychotherapies (American Psychological Association, 2019). While the efficacy of antidepressants in preventing relapse is well-established, approximately 40% of patients experience recurrence after discontinuing treatment (Kato et al., 2021). Due to the lack of clear guidelines on optimal treatment duration, some have suggested lifelong maintenance therapy. However, despite their relatively low side-effect profile, long-term antidepressant use is often reported as distressing by up to half of patients (Cascade et al., 2009).

Therefore, it is essential to identify predictive markers that can guide clinicians in deciding when it is safe to discontinue medication without increasing the risk of relapse. A recent meta-analysis conducted by our group found that demographic and clinical variables such as age, sex, or treatment resistance failed to predict recurrence (Arikan et al., 2023). Consequently, the focus has shifted to biological, electrophysiological, and genetic markers.

Objective The primary purpose (objective) of this study is to investigate whether various biological indicators provide sufficient metrics for discontinuing treatment in patients diagnosed with Major Depressive Disorder (MDD).

Study Design

The study design is described as a hybrid cohort study that integrates both retrospective and prospective data. It also incorporates an analysis strategy consistent with an unmatched case-control study methodology for sample size calculation and comparison against a Healthy Control group.

This study will enroll individuals diagnosed with MDD who respond to antidepressant treatment. Participants whose remission is maintained for 6-12 months will undergo a tapered discontinuation of their medication. They will be monitored monthly for 6-12 months following the discontinuation.

I. Study Overview and Objectives The core purpose of this research is to identify a set of multimodal biomarkers capable of predicting relapse in Major Depressive Disorder (MDD). The study is designed to answer the fundamental clinical question: "Even when a patient feels better, are they biologically recovered?" The project aims to develop a predictive algorithm that can inform clinicians on whether to continue or discontinue antidepressant medication based on objective biological data, rather than relying solely on clinical symptom assessments.

The study utilizes a hybrid cohort design, integrating retrospective data from patients with known clinical histories and prospective data from a newly recruited cohort followed over time.

II. Experimental Design and Cohorts The study is structured around three distinct participant groups to enable comprehensive comparisons.

* Group A (Retrospective / Known Phenotype): This group consists of patients with a confirmed history of either a single depressive episode or recurrent depression. Data for this group is collected at a single time point (Baseline/T0).
* Group B (Prospective / Follow-up): This cohort includes patients whose long-term outcome is unknown at the start of the study. They are enrolled, treated, and monitored over time. At the study's conclusion, they will be retrospectively categorized as "Relapsers" or "Non-Relapsers (in Remission)."
* Group C (Healthy Control): This group is composed of individuals with no history of psychiatric illness. Data is collected at a single time point to establish a healthy baseline for all biomarkers.

III. Measurement and Follow-up Timeline (Prospective Group B) The prospective cohort undergoes a series of comprehensive assessments at four key time points.

Time Point Description Measurements Taken T0 Baseline: Assessment before the initiation of antidepressant medication. All parameters measured: EEG, P300, REM, Genotype, Epigenetic i.e., Methylation, messenger Ribonucleic Acid (mRNA) expression, small ribonucleic acid (sRNA), Quality of Life (WHOQOL-BREDF) Scale, Mini Mental State Examination, Hamilton Depression Rating Scale (HDRS-17), Depression and Anxiety Stress Scale (DASS-21) T1 Early Response (4-8 weeks): An initial evaluation of treatment effect. EEG and P300 and clinical scales, i.e, HDRS-17, DASS-21 T2 Treatment Discontinuation: After a minimum of 6 months of treatment and achieving clinical remission treatment medication reduced gradually and all the measurements repeated again EEG, p300, REM, mRNA-sRNA expression, methylation, WHOQOL-BREF, HDRS-17, DASS-21 T3 End of Follow-up: The final assessment after 6 months without medication to determine relapse status. All the parameters at T2 repeated.

IV. Core Analytical Hypotheses The statistical analysis is organized into three distinct sections, each designed to test a specific set of hypotheses.

A. Baseline "Trait" Marker Identification This analysis seeks to identify stable, pre-existing biological markers that differentiate individuals with a vulnerability to recurrent depression from those who experience a single episode and from healthy controls.

* Data Pool: Combines all data from the retrospective Group A and the baseline (T0) data from the prospective Group B.
* Methodology:

  * ANOVA / Kruskal-Wallis: To compare continuous biomarker data across three groups: Recurrent, Non-Recurrent, and Healthy Controls.
  * Chi-Square Test: To analyze the relationship between categorical genetic data (SNPs) and relapse status.
* Expected Outcome: The Recurrent Depression group is expected to show biomarker profiles that are significantly different from the Healthy Control group. The Non-Recurrent group is hypothesized to fall somewhere between the Recurrent and Healthy Control groups, or to be similar to the healthy baseline.

B. Longitudinal Analysis of Biological Normalization This is the most critical component of the study, designed to test whether biological recovery aligns with clinical recovery. The central question is, "Does the biology of patients who will relapse look different from those who won't, at the moment medication is stopped?"

* Data Pool: Exclusively uses the longitudinal data from the prospective Group B (T0, T2, T3).
* Methodology: Repeated Measures ANOVA or Linear Mixed Models (LMM) will be used to analyze changes over time. The key statistical target is a significant "Group x Time" interaction effect.
* Hypothesized Scenarios:

  1. Non-Relapsing Group: Biomarkers that are abnormal at baseline (T0) are expected to normalize by the time of medication cessation (T2), becoming statistically indistinguishable from the Healthy Control group.
  2. Relapsing Group: Despite achieving clinical remission, this group's biomarkers are expected to remain abnormal at T2. The biological dysfunction will persist, indicating an incomplete recovery that predisposes them to relapse.

C. Early Treatment Response as a Predictor This analysis aims to determine if very early changes in brain activity can predict the final outcome months later.

* Data Pool: Uses T0 and T1 data (EEG/P300/HDRS-17/DASS-21) from Group B.
* Methodology: The percentage of change in measurements from T0 to T1 will be calculated. This "delta" value will then be tested for its ability to predict relapse status at T3 using point-biserial correlation or logistic regression.

The Clinical Decision Support Algorithm The final and most translational output of the study is the development of a predictive model to guide clinical practice.

* Methodology: Receiver Operating Characteristic (ROC) curve analysis will be performed.
* Process:

  1. Creation of a Normalization Index (NI): For each patient in Group B, a score will be calculated at T2 that quantifies how much their key biomarkers deviate from the healthy control average (e.g., as a Z-score).
  2. Prediction Test: The NI and other biomarker values from T2 will be used to predict the actual relapse outcome observed at T3.
  3. Performance Evaluation: The Area Under the Curve (AUC) will be calculated to measure the model's predictive accuracy. An AUC value above 0.80 is considered excellent.
  4. Cut-off Value Determination: The analysis will identify a specific biomarker threshold (a "cut-off" point) that provides the optimal balance of sensitivity and specificity for predicting relapse.
* Example Clinical Recommendation: "Based on the model, patients whose P300 latency remains above 320ms or whose specific mRNA expression is below value 'X' at the time of planned medication discontinuation have an 85% risk of relapse. It is recommended that these patients continue treatment, even if they report feeling well." V. Anticipated Conclusions and Clinical Impact

Upon completion, this study is positioned to make several powerful and field-advancing claims:

1. Identification: "The phenotype of relapsing depression is distinguishable from single-episode depression at baseline through a distinct profile of P300 amplitude deficits and specific RNA expression patterns."
2. Mechanism: "While antidepressant treatment can resolve clinical symptoms within six months, the underlying electrophysiological dysfunctions-a form of 'biological scar'-persist in the group that is destined to relapse."
3. Clinical Recommendation: "The decision to terminate antidepressant therapy should not be based solely on clinical remission as measured by scales like Hamilton. It must be guided by evidence of biological normalization, as determined by biomarker values at the point of remission."

Healthy Control Recruitment

Healthy controls will be recruited from various departments of a large corporate organization. Following informed consent, each participant will undergo psychiatric interviews conducted by board-certified psychiatrists using the Structural Clinical Interview for DSM-5 (SCID-5) and a sociodemographic questionnaire. Interview results will not be disclosed to participants. Subsequent assessments will include resting-state qEEG, event-related potentials (P300), overnight sleep EEG, and blood sampling for genetic analysis. Devices and protocols will match those used in the depression group to ensure consistency.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients
* For patients, satisfying Major Depressive Disorder for Diagnostic and Statistical Manual of Mental Disorders (DSM-5-TR)
* Drug-free for at least 1-week

Exclusion Criteria:

* Any neurological and psychiatric comorbid conditions
* Hearing loss
* Physical diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who get diagnosed with major depressive disorders according to DSM-IV or DSM-V
Sampling Method: Non-Probability Sample
Enrollment: 204 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Relapse rate | From the discontinuation of antidepressant treatment to the first relapse within 6-12 months.
  The number of person relapsed, which is evaluated by Hamilton Depression Rating Scale, after discontinuation of antidepressant treatment.

SECONDARY OUTCOMES:
Severity of Depression - Baseline (T0) | Baseline - T0: Before the start of antidepressant medication.
  Hamilton Depression Rating Scale the 17-item form will be used in the present study. Some items are scored from 0 to 4, some from 0 to 2, and some from 0 to 3. The maximum total score is 53; scores ≥29 indicate severe depression, 16-28 moderate, 8-15 mild, and 0-7 no depression.
Severity of Depression - Treatment Response (T1) | T1: 4-8 weeks after the start of antidepressant treatment (T0)
  Hamilton Depression Rating Scale the 17-item form will be used in the present study. Some items are scored from 0 to 4, some from 0 to 2, and some from 0 to 3. The maximum total score is 53; scores ≥29 indicate severe depression, 16-28 moderate, 8-15 mild, and 0-7 no depression
Severity of Depression - End of Treatment (T2) | T2: 6-12 months after the start of antidepressant medication(T0).
  Hamilton Depression Rating Scale the 17-item form will be used in the present study. Some items are scored from 0 to 4, some from 0 to 2, and some from 0 to 3. The maximum total score is 53; scores ≥29 indicate severe depression, 16-28 moderate, 8-15 mild, and 0-7 no depression
Severity of Depression - End of Study (T3) | T3: 6-12 months after the discontinuation of treatment(T2)
  Hamilton Depression Rating Scale the 17-item form will be used in the present study. Some items are scored from 0 to 4, some from 0 to 2, and some from 0 to 3. The maximum total score is 53; scores ≥29 indicate severe depression, 16-28 moderate, 8-15 mild, and 0-7 no depression.
QEEG absolute power- Baseline (T0) | Baseline (Day 0) - T0 (Patients): Before the start of antidepressant medication. Baseline (Day 0) - T0 (Controls): For the control group, this assessment is conducted at the end of initial psychiatric evaluation to establish baseline measurements.
  The absolute power in 6 main frequency bands (delta, theta, alpha, beta, high beta, gamma) for both patient and control group
QEEG absolute power at Treatment Response (T1) | T1: 4-8 weeks after the start of antidepressant treatment (T0)
  The absolute power in 6 main frequency bands (delta, theta, alpha, beta, high beta, gamma) for patient group.
QEEG absolute power - End of Treatment (T2) | T2: 6-12 months after the start of treatment (T0)
  The absolute power in 6 main frequency bands (delta, theta, alpha, beta, high beta, gamma)
QEEG absolute power - Last Relapse Control - End of the Study (T3) | T3: 6-12 months after the discontinuation of treatment(T2)
  The absolute power in 6 main frequency bands (delta, theta, alpha, beta, high beta, gamma)
P300 amplitude - Baseline (T0) | Baseline (Day 0) - T0 (Patients): Before the start of antidepressant medication. Baseline (Day 0) - T0 (Controls): For the control group, this assessment is conducted at the end of initial psychiatric evaluation to establish baseline measurements.
  The P300 amplitude in auditory oddball paradigm
P300 amplitude at Treatment Response (T1) | T1: 4-8 weeks after the start of antidepressant treatment (T0)
  The P300 amplitude in auditory oddball paradigm.
P300 amplitude- End of Treatment (T2) | T2: 6-12 months after the start of treatment (T0)
  The P300 amplitude in auditory oddball paradigm, for patients only
P300 amplitude- Last Relapse Control - End of the Study (T3) | T3: 6-12 months after the discontinuation of treatment(T2)
  The P300 amplitude in auditory oddball paradigm.
REM latency - Baseline (T0) | Baseline (Day 0) - T0 (Patients): Before the start of antidepressant medication. Baseline (Day 0) - T0 (Controls): For the control group, this assessment is conducted at the end of initial psychiatric evaluation to establish baseline measurements.
  Time until first REM period measured at sleep EEG, for both patients and healthy controls.
REM latency - End of Treatment (T2) | T2: 6-12 months after the start of treatment (T0)
  Time until first REM period measured at sleep EEG.
REM Latency Last Relapse Control - End of the Study (T3) | T3: 6-12 months after the end of treatment (T2)
  Time until first Rapid Eye Movement (REM) period measured at sleep Electroencephalography (EEG).
DNA Genome Analysis - Baseline (T0) | Baseline (Day 0) - T0 (Patients): Before the start of antidepressant medication. Baseline (Day 0) - T0 (Controls): For the control group, this assessment is conducted at the end of initial psychiatric evaluation to establish baseline measurements.
  Genotype analysis for depression related genes and pharmacogenetic analysis
RNA Sequencing - Baseline (T0) | Baseline (Day 0) - T0 (Patients): Before the start of antidepressant medication. Baseline (Day 0) - T0 (Controls): For the control group, this assessment is conducted at the end of initial psychiatric evaluation to establish baseline measurements.
  Transcriptome sequencing aims to identify all RNA molecules expressed in a given cell population at a specific time.
RNA Sequencing - End of Treatment (T2) | T2: 6-12 months after the start of antidepressant treatment (T0)
  Transcriptome sequencing aims to identify all RNA molecules expressed in a given cell population at a specific time.
RNA Sequencing - End of Study (T3) | T3: 6-12 months after the end of treatment (T2)
  Transcriptome sequencing aims to identify all RNA molecules expressed in a given cell population at a specific time.
Micro RNA Sequencing - Baseline (T0) | Baseline (Day 0) - T0 (Patients): Before the start of antidepressant medication. Baseline (Day 0) - T0 (Controls): For the control group, this assessment is conducted at the end of initial psychiatric evaluation to establish baseline measurements.
  The human genome contains short non-coding Ribo Nucleic Acid (RNA)molecules, including microRNAs These regulate various physiological and pathological processes within the cell. They control gene expression levels by degrading their target RNAs or by suppressing protein synthesis.
Micro RNA Sequencing - End of Treatment (T2) | T2: 6-12 months after the start of antidepressant treatment (T0)
  The human genome contains short non-coding Ribo Nucleic Acid (RNA)molecules, including microRNAs These regulate various physiological and pathological processes within the cell. They control gene expression levels by degrading their target RNAs or by suppressing protein synthesis.
Micro RNA Sequencing - End of Study (T3) | T3: 6-12 months after the end of treatment (T2)
  The human genome contains short non-coding Ribo Nucleic Acid (RNA)molecules, including microRNAs These regulate various physiological and pathological processes within the cell. They control gene expression levels by degrading their target RNAs or by suppressing protein synthesis.
DNA Methylation - Baseline (T0) | Baseline (Day 0) - T0 (Patients): Before the start of antidepressant medication. Baseline (Day 0) - T0 (Controls): For the control group, this assessment is conducted at the end of initial psychiatric evaluation to establish baseline measurements.
  Genome-wide DNA methylation profiles obtained by long-read whole-genome sequencing . This sequencing measures the kinetics of DNA polymerase during sequencing, it directly detect base modifications, including 5-methylcytosine (5mC), without the need for bisulfite conversion.
DNA Methylation - End of Treatment (T2) | T2: 6-12 months after the start of antidepressant treatment (T0)
  Genome-wide DNA methylation profiles obtained by long-read whole-genome sequencing . This sequencing measures the kinetics of DNA polymerase during sequencing, it directly detect base modifications, including 5-methylcytosine (5mC), without the need for bisulfite conversion.
DNA Methylation - End of Study (T3) | T3: 6-12 months after the end of treatment (T2)
  Genome-wide DNA methylation profiles obtained by long-read whole-genome sequencing . This sequencing measures the kinetics of DNA polymerase during sequencing, it directly detect base modifications, including 5-methylcytosine (5mC), without the need for bisulfite conversion.
DNA Length - Baseline (T0) | Baseline (Day 0) - T0 (Patients): Before the start of antidepressant medication. Baseline (Day 0) - T0 (Controls): For the control group, this assessment is conducted at the end of initial psychiatric evaluation to establish baseline measurements.
  PacBio's HiFi sequencing provides high-fidelity long reads, enabling the measurement and mapping of DNA sequences that span thousands of base pairs. This is particularly useful for spanning repetitive regions where the exact length of the DNA is critical.
DNA Length - End of Treatment (T2) | T2: 6-12 months after the start of antidepressant treatment (T0)
  PacBio's HiFi sequencing provides high-fidelity long reads, enabling the measurement and mapping of DNA sequences that span thousands of base pairs. This is particularly useful for spanning repetitive regions where the exact length of the DNA is critical.
DNA Length - End of Study (T3) | T3: 6-12 months after the end of treatment (T2)
  PacBio's HiFi sequencing provides high-fidelity long reads, enabling the measurement and mapping of DNA sequences that span thousands of base pairs. This is particularly useful for spanning repetitive regions where the exact length of the DNA is critical.

OTHER OUTCOMES:
Anxiety Level at Baseline (T0) | Baseline - T0: Before the start of antidepressant medication.
  The Hamilton Anxiety Rating Scale developed by Max Hamilton consisting of 14 items, each scored from 0 to 4. The maximum total score is 56; scores ≥31 indicate severe anxiety, 25-30 moderate to severe, 18-24 mild to moderate, and ≤17 mild anxiety.
Anxiety Level at Treatment Response(T1) | T1: 4-8 weeks after the start of antidepressant treatment (T0)
  The Hamilton Anxiety Rating Scale developed by Max Hamilton consisting of 14 items, each scored from 0 to 4. The maximum total score is 56; scores ≥31 indicate severe anxiety, 25-30 moderate to severe, 18-24 mild to moderate, and ≤17 mild anxiety.
Anxiety level - End of Treatment (T2) | T2: 6-12 months after the start of antidepressant medication (T0)
  The Hamilton Anxiety Rating Scale developed by Max Hamilton consisting of 14 items, each scored from 0 to 4. The maximum total score is 56; scores ≥31 indicate severe anxiety, 25-30 moderate to severe, 18-24 mild to moderate, and ≤17 mild anxiety.
Anxiety Level - End of Study (T3) | T3: 6-12 months after the discontinuation of treatment(T2)
  The Hamilton Anxiety Rating Scale developed by Max Hamilton consisting of 14 items, each scored from 0 to 4. The maximum total score is 56; scores ≥31 indicate severe anxiety, 25-30 moderate to severe, 18-24 mild to moderate, and ≤17 mild anxiety.
Stress Level at Baseline (T0) | Baseline - T0: Before the start of antidepressant medicaiton.
  Twenty one item Depression and Anxiety Stress Scale, developed by Peter and Sydney Lovibond (1995), assesses depression, anxiety, and stress severity over the past week in three seperate subscale, with 7 items per subscale scored from 0 to 3. Each subscale has a raw score range of 0-21, Higher scores indicate greater symptom severity and are classified from normal to extremely severe, reflecting symptom intensity rather than a clinical diagnosis.
Stress Level at Treatment Response (T1) | T1: 4-8 weeks after start of antidepressant medication(T0)
  Twenty one item Depression and Anxiety Stress Scale, developed by Peter and Sydney Lovibond (1995), assesses depression, anxiety, and stress severity over the past week in three seperate subscale, with 7 items per subscale scored from 0 to 3. Each subscale has a raw score range of 0-21, Higher scores indicate greater symptom severity and are classified from normal to extremely severe, reflecting symptom intensity rather than a clinical diagnosis.
Stress Level at End of Treatment (T2) | T2: 6-12 months after the start of antidepressant treatment (T0)
  Twenty one item Depression and Anxiety Stress Scale, developed by Peter and Sydney Lovibond (1995), assesses depression, anxiety, and stress severity over the past week in three seperate subscale, with 7 items per subscale scored from 0 to 3. Each subscale has a raw score range of 0-21, Higher scores indicate greater symptom severity and are classified from normal to extremely severe, reflecting symptom intensity rather than a clinical diagnosis.
Stress Level at End of Study (T3) | T3: 6-12 months after the discontinuation of treatment(T2)
  Twenty one item Depression and Anxiety Stress Scale, developed by Peter and Sydney Lovibond (1995), assesses depression, anxiety, and stress severity over the past week in three seperate subscale, with 7 items per subscale scored from 0 to 3. Each subscale has a raw score range of 0-21, Higher scores indicate greater symptom severity and are classified from normal to extremely severe, reflecting symptom intensity rather than a clinical diagnosis.
Quality of Life at Baseline (T0) | Baseline - T0: Before the start of antidepressant medication.
  The World Health Organisation Quality of Life Short Scale is a self-report quality of life scale developed by the World Health Organization. It consists of 26 items forming four domains: Physical Health (7 items), Psychological Health (6 items), Social Relationships (3 items), and Environment (8 items), plus two general items assessing overall quality of life and general health. Items are rated on a 5-point Likert scale; raw domain scores are transformed to a 0-100 scale, where higher scores indicate better quality of life, with 100 representing the maximum possible score in each domain.
Quality of Life at End of Treatment (T2) | T2: 6-12 months after the start of antidepressant treatment (T0)
  The World Health Organisation Quality of Life Short Scale is a self-report quality of life scale developed by the World Health Organization. It consists of 26 items forming four domains: Physical Health (7 items), Psychological Health (6 items), Social Relationships (3 items), and Environment (8 items), plus two general items assessing overall quality of life and general health. Items are rated on a 5-point Likert scale; raw domain scores are transformed to a 0-100 scale, where higher scores indicate better quality of life, with 100 representing the maximum possible score in each domain.
Quality of Life at End of Treatment (T3) | T3: 6-12 months after the discontinuation of treatment(T2)
  The World Health Organisation Quality of Life Short Scale is a self-report quality of life scale developed by the World Health Organization. It consists of 26 items forming four domains: Physical Health (7 items), Psychological Health (6 items), Social Relationships (3 items), and Environment (8 items), plus two general items assessing overall quality of life and general health. Items are rated on a 5-point Likert scale; raw domain scores are transformed to a 0-100 scale, where higher scores indicate better quality of life, with 100 representing the maximum possible score in each domain.
Magnetic Resonance Imaging combined with Diffusion Tensor Imaging measurement at Baseline (T0) | Baseline (Day 0) - T0 (Patients): Before the start of antidepressant medication. Baseline (Day 0) - T0 (Controls): For the control group, this assessment is conducted at the end of initial psychiatric evaluation to establish baseline measurements.
  Magnetic Resonance Imaging combined with Diffusion Tensor Imaging, for both patients and controls
Magnetic Resonance Imaging combined with Diffusion Tensor Imaging measurement at the end of study (T3) | T3: 6-12 months after the discontinuation of treatment (T2)
  Magnetic Resonance Imaging combined with Diffusion Tensor Imaging, for patients only.
Mental State - Baseline (T0) | Baseline - T0: Before the start of antidepressant medication.
  The Mini-Mental State Examination (MMSE) is a brief clinician-administered cognitive screening tool developed by Folstein, Folstein, and McHugh (1975). It consists of 30 items assessing orientation, registration, attention and calculation, recall, language, and visuospatial abilities, with a total score range of 0-30, where higher scores indicate better cognitive functioning; scores below 24 are commonly considered suggestive of cognitive impairment, depending on age and education.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Kemal Arıkan, Prof., Principal Investigator — Kemal Arikan Psychiatry Clinic
Locations (1):
- Prof. Dr. Kemal Arıkan's Psychiatry Clinic, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the primary and secondary outcome results will be shared. This includes electrophysiological (qEEG, P300, REM latency), MRI, genomic (Single Nucleotid Variations, Copy Number Variations, long-read structural variants), transcriptomic, small RNA, and methylation/genotyping data. Only fully de-identified datasets and associated data dictionaries will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be made available 12 months after publication of the primary study results and will remain available for at least 5 years thereafter. Supporting documents (protocol, Statistical Analysis Plan, Informed Consent Form, analytical code) will be released at the same time as the de-identified IPD. Long-term archiving beyond 5 years will be maintained depending on repository policies.
Access Criteria: Access will be provided to qualified researchers for scientifically sound proposals. Requests must include a study protocol, research objectives, and ethics approval from the requester's institution. All requests will be reviewed by an independent data access committee. Approved researchers must sign a Data Use Agreement. Access will be provided through a secure repository, and only de-identified data will be shared. Contact for requests: mkarikan46@gmail.com

REFERENCES:
- [Background] Arikan MK, Ilhan R, Pogarell O, Metin B. When to stop medication in unipolar depression: A systematic review and a meta-analysis of randomized controlled trials. J Affect Disord. 2023 Mar 15;325:7-13. doi: 10.1016/j.jad.2023.01.024. Epub 2023 Jan 6. PMID 36623560
- [Background] Arikan MK, Uysal O, Gica S, Orhan O, Ilhan R, Esmeray MT, Bakay H, Metin B, Pogarell O, Turan S. REM parameters in drug-free major depressive disorder: A systematic review and meta-analysis. Sleep Med Rev. 2024 Feb;73:101876. doi: 10.1016/j.smrv.2023.101876. Epub 2023 Nov 20. PMID 37995418
- [Background] Arikan MK, Ilhan R, Orhan O, Esmeray MT, Turan S, Gica S, Bakay H, Pogarell O, Tarhan KN, Metin B. P300 parameters in major depressive disorder: A systematic review and meta-analysis. World J Biol Psychiatry. 2024 Apr;25(4):255-266. doi: 10.1080/15622975.2024.2321554. Epub 2024 May 1. PMID 38493361
- [Background] Arikan MK, Ilhan R. Gamma-band qEEG biomarkers as trait indicators in depression. J Affect Disord. 2026 Jan 15;393(Pt A):120287. doi: 10.1016/j.jad.2025.120287. Epub 2025 Sep 11. PMID 40945766
- [Background] Arikan MK, Ilhan R. State-Dependent qEEG Biomarkers in Depression. Clin EEG Neurosci. 2026 Jan;57(1):17-32. doi: 10.1177/15500594251384430. Epub 2025 Oct 7. PMID 41055949

DOCUMENTS (3):
  • Study Protocol (2025-12-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT07328373/Prot_000.pdf
  • Statistical Analysis Plan (2025-12-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT07328373/SAP_001.pdf
  • Informed Consent Form (2025-12-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT07328373/ICF_002.pdf